CLINICAL TRIAL: NCT04642391
Title: Defining the Mechanisms Underlying Adrenal Dysfunction in Cirrhosis and Its Prognostic Significance
Brief Title: Defining the Mechanisms Underlying Adrenal Insufficiency in Cirrhosis
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: American Association for the Study of Liver Diseases (Other)
Responsible Party: Principal Investigator, Brian Wentworth, MD, Assistant Professor Medicine, University of Virginia
Other Study IDs: HSR200392
Record Dates: First submitted 2020-11-17; First posted 2020-11-24 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Cirrhosis; Adrenal Insufficiency
MeSH Terms: conditions — Fibrosis; Adrenal Insufficiency | interventions — Cosyntropin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RAI: Subjects will be diagnosed with relative adrenal insufficiency as determined by administration of a standard-dose ACTH stimulation test (0.25mg Cosyntropin) and an increase in serum total cortisol <9mcg/dL.
  Interventions: Drug: Cosyntropin
- Non-RAI: Subjects will have not have relative adrenal insufficiency as determined by administration of a standard-dose ACTH stimulation test (0.25mg Cosyntropin) and an increase in serum total cortisol >= 9mcg/dL.
  Interventions: Drug: Cosyntropin

INTERVENTIONS:
Drug: Cosyntropin — Administer 0.25mg Cosyntropin to determine adrenal sufficiency vs. insufficiency in patients with decompensated cirrhosis

SUMMARY:
This study aims to define the prevalence and potential pathophysiologic mechanisms underlying relative adrenal insufficiency (RAI) in outpatients with decompensated cirrhosis. Patients will be followed prospectively for up to two years to determine incidence of RAI, whether RAI represents a permanent or dynamic physiologic state in cirrhosis, and to determine whether RAI in this setting is associated with important clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18y
* Diagnosis of cirrhosis by biopsy or compatible clinical picture
* Experienced at least one portal decompensating event in the past and currently have a Child-Pugh B or C classification

Exclusion Criteria:

* Pregnant women
* Prisoners
* Not been treated with medication known to affect the adrenal axis within the past 4 weeks (oral or IV steroids, ketoconazole, etomidate)
* Hospitalized at time of enrollment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Decompensated cirrhosis (cirrhosis + at least 1 clinically-significant decompensation including ascites/hepatic hydrothorax, spontaneous bacterial peritonitis, variceal bleed, hepatic encephalopathy)
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
RAI prevalence | 1 year
Baseline Cholesterol Esterification Percentage | baseline
6 month Cholesterol Esterification Percentage | 6 months
12 month Cholesterol Esterification Percentage | 12 months
18 month Cholesterol Esterification Percentage | 18 months
24 month Cholesterol Esterification Percentage | 24 months
Baseline 17-OH Progesterone Level | baseline
6 month 17-OH Progesterone Level | 6 month
12 month 17-OH Progesterone Level | 12 months
18 month 17-OH Progesterone Level | 18 months
24 month 17-OH Progesterone Level | 24 months
Baseline ACTH level | baseline
6 month ACTH level | 6 months
12 month ACTH level | 12 months
18 month ACTH level | 18 months
24 month ACTH level | 24 months
Baseline IL-1 Level | baseline
6 month IL-1 Level | 6 months
12 month IL-1 Level | 12 months
18 month IL-1 Level | 18 months
24 month IL-1 Level | 24 months
Baseline Plasma Renin Activity | baseline
6 month Plasma Renin Activity | 6 month
12 month Plasma Renin Activity | 12 month
18 month Plasma Renin Activity | 18 month
24 month Plasma Renin Activity | 24 month
Baseline serum normetanephrine level | baseline
6 month serum normetanephrine level | 6 month
12 month serum normetanephrine level | 12 month
18 month serum normetanephrine level | 18 month
24 month serum normetanephrine level | 24 month
Baseline 11-deoxycortisol level | baseline
6 month 11-deoxycortisol level | 6 months
12 month 11-deoxycortisol level | 12 months
18 month 11-deoxycortisol level | 18 months
24 month 11-deoxycortisol level | 24 months
Baseline HDL level | baseline
6 month HDL level | 6 months
12 month HDL level | 12 months
18 month HDL level | 18 months
24 month HDL level | 24 months
Baseline IL-6 level | baseline
6 month IL-6 level | 6 months
12 month IL-6 level | 12 months
18 month IL-6 level | 18 months
24 month IL-6 level | 24 months
Baseline IL-10 level | baseline
6 month IL-10 level | 6 months
12 month IL-10 level | 12 months
18 month IL-10 level | 18 months
24 month IL-10 level | 24 months
Baseline TNFa level | baseline
6 month TNFa level | 6 months
12 month TNFa level | 12 months
18 month TNFa level | 18 months
24 month TNFa level | 24 months

SECONDARY OUTCOMES:
Annualized Incidence of RAI | over two years
30-day transplant-free survival | 30 days
90-day transplant-free survival | 90 days
6-month transplant-free survival | 6 months
1 year transplant-free survival | 1 year
2 year transplant-free survival | 2 years
30 day new or worsened portal hypertensive decompensation | 30 days
90 day new or worsened portal hypertensive decompensation | 90 days
6 month new or worsened portal hypertensive decompensation | 6 months
1 year new or worsened portal hypertensive decompensation | 1 year
2 year new or worsened portal hypertensive decompensation | 2 years
30 day unplanned hospitalization | 30 days
90 day unplanned hospitalization | 90 days
6 month unplanned hospitalization | 6 month
1 year unplanned hospitalization | 1 year
2 year unplanned hospitalization | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No